CLINICAL TRIAL: NCT04382352
Title: Experimental Study on the Safety, Tolerability, Pharmacokinetics and Efficacy of B002 in the Treatment of HER2-positive Recurrent or Metastatic Breast Cancer.
Brief Title: B002 in Patients With HER2-positive Breast Cancer
Acronym: B002-101
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Pharmaceuticals Holding Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B002-101
Record Dates: First submitted 2020-04-29; First posted 2020-05-11 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2022-10

CONDITIONS: Recurrent Breast Cancer; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Biological Products; Injections

STUDY DESIGN:
Intervention Model Description: Test staging: Phase I Design Type: Single Arm Test This study was a preliminary study of stage Ia, openness, dose escalation, pharmacokinetics, and efficacy.
  To assess safety and tolerability in HER2-positive recurrent or metastatic breast cancer subjects, to determine dose-limiting toxicity (DLT) and to explore maximum tolerated dose (MTD); to evaluate pharmacokinetic characteristics, immunization Originality and preliminary exploration of efficacy.
  The study was divided into the main trial period and the extended trial period. The subject trial completed the enrollment and DLT observations of all evaluable DLT subjects for the dose climbing phase; the PK expansion phase completed the enrollment required PK sample collection for the enrolled subjects.
  The extension test is the completion of the subject test and the subject continues to take the drug to the stage of progression of the disease or intolerance.
  Blind method: open Test range: Domestic test
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Humanized Anti-HER2 Monoclonal Antibody Compound for Injection (Experimental): Registration number: CTR20181455 Indications: HER2-positive recurrent or metastatic breast cancer Experimental popular topic: Phase Ia clinical study of recombinant anti-HER2 humanized monoclonal antibody composition
  Interventions: Biological: Humanized Anti-HER2 Monoclonal Antibody Compound for Injection .R&D code: B002.

INTERVENTIONS:
Biological: Humanized Anti-HER2 Monoclonal Antibody Compound for Injection .R&D code: B002. — Usage: intravenous infusion; B002, doses 2, 6, 12, 16, 20 mg / kg, intravenous drip. The infusion time was 120 ± 10 minutes for the first time; if the patient was tolerated, the follow-up time was adjusted to 60 ± 10 minutes. Pre-treatment was performed using phenergan (25 mg, intramuscular) within 30 minutes prior to each study drug infusion. The dosing cycle is administered once every 3 weeks for one cycle and can be administered continuously until the disease progresses or is intolerable.
  Other Names: Biological Products; Humanized Anti-HER2 Monoclonal Antibody Compound for Injection

SUMMARY:
To assess the safety and tolerability characteristics of B002 in patients with HER2-positive recurrent or metastatic breast cancer. The dose-limiting toxicity (DLT) was assessed and the maximum tolerated dose (MTD) was explored.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old ≤ age ≤ 70 years old, female;
* BMI 18 ~ 32 kg / m2, including both ends;
* Histological or cytologically confirmed recurrent or metastatic breast cancer. According to RECIST v 1.1, patients with measurable and/or unmeasurable lesions:

  1. Patients with bone metastases, as long as the bone metastases have never received radiotherapy, and the primary tumor tumours are available for HER2 detection and Biomarker analysis, which can be enrolled;
  2. Patients with local recurrence and unsuitable for radical mastectomy;
  3. For bilateral breast cancer, and bilateral HER2 expression is inconsistent, the metastases should be confirmed to be HER2 positive;
* Anti-HER2 treatment failure for recurrent or metastatic disease;
* A retrograde or metastatic breast cancer diagnosed as HER2 positive (FISH positive and / or IHC 3+) by the Department of Pathology diagnosis;
* The left ventricular ejection fraction (LVEF) was detected by echocardiography (ECHO) ≥50% in the baseline period (28 days before the start of the trial);
* ECOG physical state (PS) is 0-1 points;
* Expected to survive for more than 3 months;
* Female patients of childbearing age, patients and/or their partners should agree to use a highly effective non-hormonal contraceptive method or two effective non-hormonal contraceptive methods. Continue to use the appropriate contraceptive measures during the study period and at least 6 months after the last dose;
* Understand and voluntarily sign the informed consent form.

Exclusion Criteria:

* In the screening examination, the blood concentration of patients who have used pertuzumab in the past is ≥5μg/ml;
* In the screening examination, the blood concentration of patients who have used trastuzumab in the past is ≥5μg/ml;
* Known to be allergic to the study drug or its components;
* Subjects with a history of contrast allergies;
* There is clinical or radiological evidence of a central nervous system (CNS) metastasis. For patients with clinically suspected CNS metastases, enhanced CT or enhanced MRI must be performed within the first 28 days of randomization to exclude CNS metastasis;
* Hematological toxicity caused by previous treatment CTCAE ≥ 2 persistence (except hemoglobin) (NCI-CTCAE version 4.03);
* There are peripheral neuropathy CTCAE ≥ 3 (first dose group, peripheral neuropathy CTCAE ≥ 2);
* A history of other malignancies in the last 5 years, except for cured cervical carcinoma in situ or basal cell carcinoma or squamous cell carcinoma of the skin;
* Uncontrolled high blood pressure (systolic blood pressure greater than 150 mmHg and / or diastolic blood pressure greater than 100 mmHg), orthostatic hypotension;
* Cardiac standard: QTc>480ms. There are factors that can cause QTc prolongation or arrhythmia such as congestive heart failure, hypokalemia, long QT syndrome (atrial fibrillation, paroxysmal supraventricular tachycardia). There are any unstable cardiovascular diseases (including the New York Heart Association NYHA cardiac function grade III or IV, congestive heart failure, unstable angina, a history of myocardial infarction within 6 months);
* LVEF <50% during the period of neoadjuvant or adjuvant therapy or prior to the end of treatment with trastuzumab or pertuzumab for injection;
* Resting dyspnea caused by complications of advanced malignancies, or other conditions requiring continuous oxygen therapy;
* There are serious, uncontrollable systemic diseases (such as clinically significant cardiovascular, pulmonary, liver and kidney, digestive or metabolic diseases; fractures);
* Experience major surgery or trauma within 28 days prior to the start of the trial, or plan for major surgery before the end of the study treatment;
* The cumulative dose of anthracycline antibiotics was assessed at baseline (within 28 days prior to the start of the trial) to meet the following criteria:

  1. doxorubicin > 360 mg/m2;
  2. epirubicin > 720 mg/m2;
  3. hydrochloric acid mitoxantrone > 120 mg/m2 and idarubicin (demethoxy daunorubicin) > 90 mg/m2;
  4. other (such as doxorubicin liposome or other anthracycline antibiotics > 360 mg / Doxorubicin equivalent dose of m2);
  5. If more than one anthracycline antibiotic is used, the cumulative dose should not exceed the equivalent dose of doxorubicin of 360 mg/m2;
* Have received any trial medication within 28 days prior to the start of the trial;
* Have received any therapeutic antibody or vaccine within 28 days prior to the start of the trial;
* Chemotherapy, endocrine therapy, and radiotherapy were administered within 28 days prior to the start of the trial;
* Intravenous infusion of antibiotics to treat infection within 14 days prior to the start of the trial;
* Daily oral glucocorticoid treatment, equivalent to a dose of >10 mg / day of methylprednisolone, except for inhaled corticosteroids;
* The presence of anti-drug antibodies against trastuzumab or pertuzumab;
* Within 7 days prior to the start of the trial, laboratory tests revealed any of the following abnormalities:

  1. Absolute count of neutral cells <1.5×109/L;
  2. Platelet count <80.0×109/L;
  3. Hemoglobin <9 g/dL;
  4. Total Bilirubin > 1.5 × normal upper limit (ULN) (unless the patient has Glibert's syndrome)
  5. AST or ALT > 2.5 × ULN
  6. Creatinine clearance (calculated using the Cockcroft_Gault formula) < 50 mL / min
  7. International normalized ratio (INR) and Activated partial thromboplastin time or partial thromboplastin time (APPT or PT) > 1.5 x ULN (unless treated for coagulation abnormalities);
* Hepatitis B surface antigen positive and HBV-DNA test ≥ lower limit of detection; hepatitis C antibody positive; HIV antibody positive;
* Pregnant or lactating women;
* Other circumstances judged by the investigator are not suitable for participation in the study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Enrollment: 23 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2022-04-26 (Actual); Study Completion 2022-04-26 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 21 days
Dose-Limiting Toxicity (DLT) | 21 days

SECONDARY OUTCOMES:
Tmax | 21 days
  Pharmacokinetics measurement
Cmax | 21 days
  Pharmacokinetics measurement
AUC | 21 days
  Pharmacokinetics measurement
Anti-drug antibody (ADA) | through study completion, an average of 2 years
Objective Remission Rate (ORR) | through study completion, an average of 2 years
  Therapeutic Efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Xichun Hu, Principal Investigator — Cancer Hospital affiliated to Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No